CLINICAL TRIAL: NCT00399542
Title: Phase 3, 12-Week, Multicenter, Double-Blind, Randomized, Efficacy and Safety Study of Lubiprostone for the Treatment of Irritable Bowel Syndrome With Constipation
Brief Title: Efficacy and Safety of Lubiprostone in Patients With Irritable Bowel Syndrome With Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sucampo Pharma Americas, LLC (Industry)
Collaborators: Sucampo Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0211SIB-0432
Record Dates: First submitted 2006-11-13; First posted 2006-11-15 (Estimated); Results first posted 2008-10-31 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2013-09

CONDITIONS: Irritable Bowel Syndrome; Constipation
Keywords: Irritable Bowel Syndrome With Constipation
MeSH Terms: conditions — Irritable Bowel Syndrome; Constipation | interventions — Lubiprostone

INTERVENTIONS:
Drug: Lubiprostone
Drug: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the efficacy and safety of administration of lubiprostone in patients with irritable bowel syndrome with constipation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Stable fiber therapy
* Normal colonoscopy/sigmoidoscopy
* Able to refrain from use of medications known to treat or associated with constipation symptoms
* Experiences abdominal discomfort/pain associated with bowel movements
* Reports decreased bowel movement frequency and/or other symptoms associated with constipation

Exclusion Criteria:

* Diarrhea-predominant or alternating (diarrhea & constipation cycling) IBS, or constipation other than that associated with IBS
* Open gastrointestinal or abdominal surgery prior to IBS onset
* Organic bowel disorder, mechanical bowel obstruction, pseudo-obstruction, unexplained weight loss or rectal bleeding
* Uncontrolled cardiovascular, liver or lung disease, neurologic or psychiatric disorder, other systemic disease, or abnormal laboratory tests per investigator discretion
* If female, is currently pregnant or nursing, or plans to become pregnant or nurse during the clinical study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 581 (Actual)
Dates: Start 2005-05; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Sucampo Pharmaceuticals, Inc.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled 05/19/05; last subject observed 08/02/06, at 65 centers across the US
Pre-assignment Details: Subjects were enrolled after an up to 4 week screening period to meet inclusion/exclusion criteria and randomized on Day 0
Groups:
- Lubiprostone: Subjects who received active drug
- Placebo: Subjects who received placebo
Period: Overall Study
Arm/Group | Lubiprostone | Placebo
Started | 387 | 194
Completed | 303 | 151
Not Completed | 84 | 43
Not completed — Adverse Event | 18 | 15
Not completed — Protocol Violation | 13 | 3
Not completed — Withdrawal by Subject | 28 | 10
Not completed — Lack of Efficacy | 18 | 8
Not completed — Lost to Follow-up | 6 | 6
Not completed — Other | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lubiprostone | Placebo | Total
Number analyzed (Participants) | 379 | 192 | 571
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (12.93) | 47.3 (13.34) | 46.1 (13.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 343 | 179 | 522
  Male | 36 | 13 | 49
Height [Mean (Standard Deviation); unit: inches] | 64.7 (3.15) | 65.0 (3.34) | 64.8 (3.21)

OUTCOME MEASURES:

1. Primary Outcome: Overall Responder Status
Description: Overall responder: monthly responder for at least 2 out of 3 months
  Monthly responder: >=Moderately relieved symptoms 4 weeks/month or Significantly relieved >= 2 weeks/month IF:
  Rescue med use did not increase; AND patient did not discontinue during the month for lack of efficacy; AND no Moderately worse or Significantly worse response in month.
Time Frame: 12 weeks
Population: Intention to treat (ITT), without Last Observational Carried Forward (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
percentage of participants | 12.1 | 5.7
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; 70.6% improvement in response with lubiprostone at 90% statistical power; Test type: Superiority or Other; p = 0.023, Cochran-Mantel-Haenszel — No adjustment; Stratified by pooled center, used to test the null hypothesis of equal rates between the 2 groups vs. the alternate hypothesis of non-equality

2. Secondary Outcome: Month 1 Spontaneous Bowel Movement Rates Change From Baseline
Description: Any bowel movement not associated with rescue medication use
Time Frame: 28 days
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: spontaneous bowel movements (SBMs)/week
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
spontaneous bowel movements (SBMs)/week | 1.55 (3.071) | 1.29 (2.934)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.391, van Elteren nonparametric test; Adjusted for center

3. Secondary Outcome: Month 1 Stool Consistency Change From Baseline
Description: 0 = Very loose (watery), 1 = Loose, 2 = Normal, 3 = Hard, 4 = Very hard (little balls)
Time Frame: 28 days
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
units on a scale | -0.47 (0.673) | -0.37 (0.582)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.151, van Elteren nonparametric test; Adjusted for center

4. Secondary Outcome: Month 1 Bowel Straining Change From Baseline
Description: 0 = Absent,1 = Mild, 2 = Moderate, 3 = Severe, and 4 = Very Severe
Time Frame: 28 days
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
units on a scale | -0.54 (0.719) | -0.42 (0.628)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.163, van Elteren nonparametric test; Adjusted for center

5. Secondary Outcome: Month 1 Constipation Severity Change From Baseline
Description: 0 = Absent, 1 = Mild, 2 = Moderate, 3 = Severe, and 4 = Very Severe
Time Frame: 28 days
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
units on a scale | -0.41 (0.606) | -0.33 (0.495)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.185, van Elteren nonparametric test; Adjusted for center

6. Secondary Outcome: Month 1 Symptom Relief
Description: * 3 = Significantly worse, -2 = Moderately worse,
  * 1 = A little bit worse, 0 = Unchanged, 1 = A little bit relieved, 2 = Moderately relieved, 3 = Significantly relieved
Time Frame: 28 days
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
units on a scale | 0.69 (1.058) | 0.60 (1.043)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.300, Cochran-Mantel-Haenszel

7. Secondary Outcome: Month 1 Responder Rate
Description: Monthly responder: >=Moderately relieved symptoms 4 weeks/month or Significantly relieved >= 2 weeks/month IF:
  Rescue med use did not increase; AND patient did not discontinue during the month for lack of efficacy; AND no Moderately worse or Significantly worse response in month.
Time Frame: 28 days
Population: ITT without LOCF
Measure: Number; unit: percentage of participants
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
percentage of participants | 9.8 | 6.8
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.303, Cochran-Mantel-Haenszel — Sequential closed testing procedures were employed; [statistical method as in outcome 1, analysis 1]

8. Secondary Outcome: Month 2 Responder Rate
Description: as for outcome 7
Time Frame: 28 days
Population: ITT without LOCF
Measure: Number; unit: percentage of participants
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
percentage of participants | 16.1 | 9.9
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.047, Cochran-Mantel-Haenszel — Sequential closed testing procedures were employed; [statistical method as in outcome 1, analysis 1]

9. Secondary Outcome: Month 3 Responder Rate
Description: as for outcome 7
Time Frame: 28 days
Population: ITT without LOCF
Measure: Number; unit: percentage of participants
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
percentage of participants | 13.5 | 5.7
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.008, Cochran-Mantel-Haenszel — Sequential closed testing procedures were employed; [statistical method as in outcome 1, analysis 1]

10. Secondary Outcome: Month 1 Abdominal Pain Change From Baseline
Description: 0 = Absent, 1 = Mild, 2 = Moderate, 3 = Severe, and 4 = Very Severe
Time Frame: 28 days
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
units on a scale | -0.32 (0.600) | -0.29 (0.450)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.663, van Elteren nonparametric test; Adjusted for center

11. Secondary Outcome: Month 2 Abdominal Pain Change From Baseline
Description: 0 = Absent, 1 = Mild, 2 = Moderate, 3 = Severe, and 4 = Very Severe
Time Frame: 28 days
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
units on a scale | -0.44 (0.707) | -0.33 (0.601)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.224, van Elteren nonparametric test; Adjusted for center

12. Secondary Outcome: Month 3 Abdominal Pain Change From Baseline
Description: 0 = Absent, 1 = Mild, 2 = Moderate, 3 = Severe, and 4 = Very Severe
Time Frame: 28 days
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
units on a scale | -0.47 (0.746) | -0.35 (0.619)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.271, van Elteren nonparametric test; Adjusted for center

13. Secondary Outcome: Month 1 Abdominal Bloating Change From Baseline
Description: 0 = Absent, 1 = Mild, 2 = Moderate, 3 = Severe, and 4 = Very Severe
Time Frame: 28 days
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
units on a scale | -0.31 (0.614) | -0.28 (0.430)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.945, van Elteren nonparametric test; Adjusted for center

14. Secondary Outcome: Month 2 Abdominal Bloating Change From Baseline
Description: 0 = Absent, 1 = Mild, 2 = Moderate, 3 = Severe, and 4 = Very Severe
Time Frame: 28 days
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
units on a scale | -0.43 (0.741) | -0.33 (0.611)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.352, van Elteren nonparametric test

15. Secondary Outcome: Month 3 Abdominal Bloating Change From Baseline
Description: 0 = Absent, 1 = Mild, 2 = Moderate, 3 = Severe, and 4 = Very Severe
Time Frame: 28 days
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
units on a scale | -0.45 (0.760) | -0.35 (0.641)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.180, van Elteren nonparametric test; Adjusted for center

16. Secondary Outcome: Month 2 Spontaneous Bowel Movement Rates Change From Baseline
Description: Any bowel movement not associated with rescue medication use
Time Frame: 28 days
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: SBMs/week
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
SBMs/week | 1.61 (3.191) | 1.39 (3.495)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.275, van Elteren nonparametric test; Adjusted for center

17. Secondary Outcome: Month 3 Spontaneous Bowel Movement Rates Change From Baseline
Description: Any bowel movement not associated with rescue medication use
Time Frame: 28 days
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: SBMs/week
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
SBMs/week | 1.43 (3.061) | 1.42 (3.584)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.722, van Elteren nonparametric test; Adjusted for center

18. Secondary Outcome: Month 2 Stool Consistency Change From Baseline
Description: 0 = Very loose (watery), 1 = Loose, 2 = Normal, 3 = Hard, 4 = Very hard (little balls)
Time Frame: 28 days
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
units on a scale | -0.50 (0.700) | -0.41 (0.724)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.177, van Elteren nonparametric test; Adjusted for center

19. Secondary Outcome: Month 3 Stool Consistency Change From Baseline
Description: 0 = Very loose (watery), 1 = Loose, 2 = Normal, 3 = Hard, 4 = Very hard (little balls)
Time Frame: 28 days
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
units on a scale | -0.49 (0.686) | -0.39 (0.748)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.082, van Elteren nonparametric test; Adjusted for center

20. Secondary Outcome: Month 2 Bowel Straining Change From Baseline
Description: 0 = Absent,1 = Mild, 2 = Moderate, 3 = Severe, and 4 = Very Severe
Time Frame: 28 days
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
units on a scale | -0.62 (0.817) | -0.50 (0.745)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.110, van Elteren nonparametric test; Adjusted for center

21. Secondary Outcome: Month 3 Bowel Straining Change From Baseline
Description: 0 = Absent,1 = Mild, 2 = Moderate, 3 = Severe, and 4 = Very Severe
Time Frame: 28 days
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
units on a scale | -0.63 (0.813) | -0.50 (0.803)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.146, van Elteren nonparametric test; Adjusted for center

22. Secondary Outcome: Month 2 Constipation Severity Change From Baseline
Description: 0 = Absent, 1 = Mild, 2 = Moderate, 3 = Severe, and 4 = Very Severe
Time Frame: 28 days
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
units on a scale | -0.51 (0.732) | -0.42 (0.664)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.373, van Elteren nonparametric test; Adjusted for center

23. Secondary Outcome: Month 3 Constipation Severity Change From Baseline
Description: 0 = Absent, 1 = Mild, 2 = Moderate, 3 = Severe, and 4 = Very Severe
Time Frame: 28 days
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
units on a scale | -0.53 (0.760) | -0.42 (0.679)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.339, van Elteren nonparametric test; Adjusted for center

24. Secondary Outcome: Month 2 Symptom Relief
Description: as for outcome 6
Time Frame: 28 days
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
units on a scale | 0.79 (1.140) | 0.55 (1.256)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.023, Cochran-Mantel-Haenszel

25. Secondary Outcome: Month 3 Symptom Relief
Description: as for outcome 6
Time Frame: 28 days
Population: ITT with LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
units on a scale | 0.75 (1.249) | 0.56 (1.222)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.073, Cochran-Mantel-Haenszel

26. Secondary Outcome: Month 3 Quality of Life Change From Baseline
Description: IBS-QOL questionnaire included 34 questions with 5 possible responses yielding the following sub-categories: dysphoria, interference with activity, body image, health worry, food avoidance, social reaction, sexual, and relationship Results range from 34 (low) to 100 (high); meaningful clinical improvement=14 point increase
Time Frame: 12 weeks
Population: ITT without LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
units on a scale | 17.3 (17.46) | 13.4 (16.26)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.062, ANCOVA; Adjusted for center

27. Secondary Outcome: Month 1 Bowel Movement Rates Change From Baseline
Time Frame: 28 days
Population: ITT, with LOCF
Measure: Mean (Standard Deviation); unit: bowel movements (BMs)/week
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
bowel movements (BMs)/week | 1.30 (2.787) | 0.87 (3.104)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.060, van Elteren nonparametric test

28. Secondary Outcome: Month 2 Bowel Movement Rates Change From Baseline
Time Frame: 28 days
Population: ITT, with LOCF
Measure: Mean (Standard Deviation); unit: BMs/week
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
BMs/week | 1.29 (2.875) | 0.95 (3.444)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.290, van Elteren nonparametric test

29. Secondary Outcome: Month 3 Bowel Movement Rates Change From Baseline
Time Frame: 28 days
Population: ITT, with LOCF
Measure: Mean (Standard Deviation); unit: BMs/week
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 379 | 192
BMs/week | 1.17 (2.757) | 0.97 (3.309)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority or Other; p = 0.495, van Elteren nonparametric test

ADVERSE EVENTS:
Arm/Group | Lubiprostone | Placebo
Serious Adverse Events (participants affected / at risk) | 2 | 2
Other Adverse Events (participants affected / at risk) | 67 | 30
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Lubiprostone | Placebo
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/384 (0) | 1/195 (1)
Cholecystitis (Hepatobiliary disorders) | 1/384 (1) | 0/195 (0)
Non-cardiac chest pain (General disorders) | 1/384 (1) | 0/195 (0)
Small intestine gangrene (Gastrointestinal disorders) | 0/384 (0) | 1/195 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0/384 (0) | 1/195 (1)
Abdominal adhesions (Gastrointestinal disorders) | 0/384 (0) | 1/195 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Lubiprostone | Placebo
Nausea (Gastrointestinal disorders) | 34/384 (34) | 11/195 (11)
Diarrhoea (Gastrointestinal disorders) | 23/384 (23) | 10/195 (10)
Headache (Nervous system disorders) | 16/384 (16) | 11/195 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No